CLINICAL TRIAL: NCT01555697
Title: Biomarker Strategies for Medication-Enhanced Cognitive Training in Schizophrenia
Acronym: Swerdlow-R34
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Neal R. Swerdlow, M.D., Ph.D., Professor, University of California, San Diego
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: NIMH-R34-MH093453-NS
Record Dates: First submitted 2012-03-13; First posted 2012-03-15 (Estimated); Results first posted 2020-08-10 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-09

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; prepulse inhibition; neurocognition; working memory; memantine; MATRICS Consensus Cognitive Battery
MeSH Terms: conditions — Schizophrenia | interventions — Memantine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Memantine/high (Active Comparator): memantine 20 mg
  Interventions: Drug: Memantine
- Placebo/high (Placebo Comparator): placebo comparator for memantine 20 mg
  Interventions: Drug: Placebo
- Memantine/low (Active Comparator): memantine 10 mg
  Interventions: Drug: Memantine
- Placebo/low (Placebo Comparator): placebo comparator for memantine 10 mg
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Memantine — Each participant receives a single pill of placebo or active drug (memantine, 10 or 20 mg) and completes about 6 hours of testing in the laboratory. One week later, that participant receives a single pill of the alternate comparator and is again tested in the laboratory. Thus, in total, each participant receives one placebo pill and one active pill, separated by one week.
  Other Names: Namenda
  Arms: Memantine/high; Memantine/low
Drug: Placebo — Each participant receives a single pill of placebo or active drug (memantine, 10 or 20 mg) and completes about 6 hours of testing in the laboratory. One week later, that participant receives a single pill of the alternate comparator and is again tested in the laboratory. Thus, in total, each participant receives one placebo pill and one active pill, separated by one week.
  Arms: Placebo/high; Placebo/low

SUMMARY:
Cognitive training is moderately effective at reducing symptoms and improving life function in schizophrenia patients. The present application develops a strategy for increasing the effectiveness of cognitive training through the use of pro-cognitive medications. Specific biomarkers will be studied that identify patients most sensitive to these pro-cognitive medications, to test the feasibility of using these biomarkers in a large clinical trial of medication-enhanced cognitive training in schizophrenia.

DETAILED DESCRIPTION:
This R34 application responds to PAR-09-173, to achieve the first goal of this FOA by supporting: "the development and/or pilot testing of new or adapted interventions." The two overarching goals of this application are: 1) to test the effects of the acute administration of the NMDA antagonist, memantine (MEM), on sensorimotor gating and working memory (WM) in schizophrenia (SZ) patients, and 2) to assess the feasibility of using MEM to predictably enhance the therapeutic benefits of cognitive training in SZ.

The pharmacotherapy of SZ has been dominated by antidopaminergic drugs with limited clinical impact. Some forms of psychosocial rehabilitation, such as cognitive training (CT), appear to effectively reduce symptoms and improve function in SZ. The premise of this application is that the benefits of CT in SZ might be enhanced by drugs that increase specific cognitive abilities, including WM, even if these pro-cognitive drugs lack clinical impact when administered without CT. The main goal of this application is to develop an innovative intervention strategy that enhances the clinical benefits of CT in SZ through administration of a pro-cognitive agent to biomarker-identified sensitive patients.

The investigators reported that a single dose of the widely used Alzheimer's disease medication, MEM (20 mg p.o.), significantly increased prepulse inhibition (PPI) of the startle reflex in healthy subjects. PPI-enhancing effects of MEM in healthy subjects are associated with: 1) increased WM; and 2) phenotypes linked to the high activity Val158Met COMT polymorphism. PPI is consistently impaired in SZ patients; lowest levels of PPI in patients are associated with: 1) poor functional outcome; and 2) the Val/Val COMT genotype. If our MEM findings in healthy subjects are reproduced in SZ patients, the investigators will detect MEM-associated improvements in PPI and WM, particularly among Val/Val patients. The investigators will then be positioned to test the hypothesis that acute PPI and WM-enhancing effects of MEM predict therapeutic benefit of MEM in SZ patients undergoing CT.

This application has two aims: Aim 1 will assess the acute effects of MEM (0 vs. 10 or 0 vs. 20 mg p.o.) in 60 SZ patients, to test the prediction that MEM will increase PPI and enhance WM in SZ patients, particularly in those characterized by low basal PPI levels and/or the Val/Val COMT genotype. Mismatch negativity and gamma band synchronization will also be assessed as potentially informative MEM-sensitive and functionally relevant biomarkers. Aim 2 will assess the feasibility of testing the therapeutic benefit of MEM as an adjunct to CT in SZ patients, and the feasibility of testing the primary hypothesis that such benefit will be predicted by increased PPI and/or WM in SZ patients after the Aim 1 single dose MEM challenge. It is predicted that subject recruitment and completion in both arms of a controlled 12-week CT trial in SZ out-patients among subjects completing Aim 1 will be appropriate for testing both the overall effectiveness of MEM as an adjunct to CT and the ability to predict this effectiveness among biomarker-identified patient subgroups.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of schizophrenia or schizoaffective disorder - depressed type

Exclusion Criteria:

* Age range,
* Current alcohol or drug abuse

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2014-07; Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Diego, San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Subjects With Schizophrenia: Placebo 1st, Then 10 mg Memantine: This is a crossover design with 2 active doses used as between-subject factors. Schizophrenia subjects in this arm receive a single pill of placebo followed by about 6 hours of testing in the laboratory. One week later, that participant receives a single 10 mg pill of memantine and is again tested in the laboratory.
- Healthy Subjects: Placebo 1st, Then 10 mg Memantine: This is a crossover design with 2 active doses used as between-subject factors. Healthy participant in this arm receive a single pill of placebo followed by about 6 hours of testing in the laboratory. One week later, that participant receives a single 10 mg pill of memantine and is again tested in the laboratory.
- Subjects With Schizophrenia: 10 mg Memantine 1st, Then Placebo: This is a crossover design with 2 active doses used as between-subject factors. Schizophrenia subjects in this arm receive a single 10 mg pill of memantine followed by about 6 hours of testing in the laboratory. One week later, that participant receives a single pill of placebo and is again tested in the laboratory.
- Healthy Subjects: 10 mg Memantine 1st, Then Placebo: This is a crossover design with 2 active doses used as between-subject factors. Healthy participants in this arm receive a single 10 mg pill of memantine followed by about 6 hours of testing in the laboratory. One week later, that participant receives a single pill of placebo and is again tested in the laboratory.
- Subjects With Schizophrenia: Placebo 1st, Then 20 mg Memantine: This is a crossover design with 2 active doses used as between-subject factors. Schizophrenia subjects in this arm receive a single pill of placebo followed by about 6 hours of testing in the laboratory. One week later, that participant receives a single 20 mg pill of memantine and is again tested in the laboratory.
- Healthy Subjects: Placebo 1st, Then 20 mg Memantine: This is a crossover design with 2 active doses used as between-subject factors. Healthy participant in this arm receive a single pill of placebo followed by about 6 hours of testing in the laboratory. One week later, that participant receives a single 20 mg pill of memantine and is again tested in the laboratory.
- Subjects With Schizophrenia: 20 mg Memantine 1st, Then Placebo: This is a crossover design with 2 active doses used as between-subject factors. Schizophrenia subjects in this arm receive a single 20 mg pill of memantine followed by about 6 hours of testing in the laboratory. One week later, that participant receives a single pill of placebo and is again tested in the laboratory.
- Healthy Subjects: 20 mg Memantine 1st, Then Placebo: This is a crossover design with 2 active doses used as between-subject factors. Healthy participants in this arm receive a single 20 mg pill of memantine followed by about 6 hours of testing in the laboratory. One week later, that participant receives a single pill of placebo and is again tested in the laboratory.
Period: Overall Study
Arm/Group | Subjects With Schizophrenia: Placebo 1st, Then 10 mg Memantine | Healthy Subjects: Placebo 1st, Then 10 mg Memantine | Subjects With Schizophrenia: 10 mg Memantine 1st, Then Placebo | Healthy Subjects: 10 mg Memantine 1st, Then Placebo | Subjects With Schizophrenia: Placebo 1st, Then 20 mg Memantine | Healthy Subjects: Placebo 1st, Then 20 mg Memantine | Subjects With Schizophrenia: 20 mg Memantine 1st, Then Placebo | Healthy Subjects: 20 mg Memantine 1st, Then Placebo
Started | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10
6 Hours Lab Testing Day 1 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10
Approx 7 Day Washout | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10
6 Hours Lab Testing Day 2 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10
Completed | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Subjects With Schizophrenia: Placebo 1st, Then 10 mg Memantine | Healthy Subjects: Placebo 1st, Then 10 mg Memantine | Subjects With Schizophrenia: 10 mg Memantine 1st, Then Placebo | Healthy Subjects: 10 mg Memantine 1st, Then Placebo | Subjects With Schizophrenia: Placebo 1st, Then 20 mg Memantine | Healthy Subjects: Placebo 1st, Then 20 mg Memantine | Subjects With Schizophrenia: 20 mg Memantine 1st, Then Placebo | Healthy Subjects: 20 mg Memantine 1st, Then Placebo | Total
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 80
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 32.4 [19 to 46] | 26.4 [20 to 43] | 39.2 [29 to 45] | 32.0 [21 to 45] | 38.9 [28 to 48] | 29.6 [21 to 36] | 35.7 [21 to 48] | 23.8 [19 to 32] | 32 [19 to 48]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 2 | 2 | 4 | 4 | 4 | 3 | 22
  Male | 8 | 9 | 8 | 8 | 6 | 6 | 6 | 7 | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 2 | 1 | 3 | 1 | 2 | 5 | 18
  Not Hispanic or Latino | 8 | 8 | 7 | 9 | 7 | 9 | 8 | 5 | 61
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3
  Asian | 2 | 4 | 0 | 0 | 0 | 4 | 3 | 3 | 16
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Black or African American | 3 | 0 | 0 | 2 | 5 | 0 | 2 | 2 | 14
  White | 3 | 5 | 8 | 7 | 4 | 5 | 3 | 3 | 38
  More than one race | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2
  Unknown or Not Reported | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 6
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 80

OUTCOME MEASURES:

1. Primary Outcome: Prepulse Inhibition
Description: Prepulse inhibition of the startle reflex is the automatic reduction in startle magnitude (assessed here by EMG of orbicularis oculi) when a startling stimulus (here a 40 ms 118 dB(A) noise burst; "PULSE") is preceded (here 10 - 120 msec) by a weak stimulus (here a 20 msec burst 16 dB over background "PREPULSE"). A %PPI metric is calculated based on the relative startle magnitude on (PREPULSE + PULSE) trials vs. PULSE alone trials. Possible maximal inhibition is 100%; there is no maximal "negative" value of inhibition. There is no clear "advantage" or "disadvantage" for lower or higher %PPI values, though on average, schizophrenia patients demonstrate lower % values compared to matched healthy subjects.
Time Frame: approx 45 minutes
Measure: Mean (Standard Error); unit: % inhibition of startle
Arm/Group | Subjects With Schizophrenia: Placebo 1st, Then 10 mg Memantine | Healthy Subjects: Placebo 1st, Then 10 mg Memantine | Subjects With Schizophrenia: 10 mg Memantine 1st, Then Placebo | Healthy Subjects: 10 mg Memantine 1st, Then Placebo | Subjects With Schizophrenia: Placebo 1st, Then 20 mg Memantine | Healthy Subjects: Placebo 1st, Then 20 mg Memantine | Subjects With Schizophrenia: 20 mg Memantine 1st, Then Placebo | Healthy Subjects: 20 mg Memantine 1st, Then Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10
% inhibition of startle
  Placebo | 30.4 (5.7) | 25.5 (8.1) | 23.7 (6.0) | 2.6 (19.2) | -1.7 (9.9) | -9.7 (33.2) | 34.2 (8.7) | 12.1 (7.3)
  Memantine | 28.9 (6.8) | 27.3 (6.5) | -0.9 (13.7) | 31.1 (8.1) | 26.1 (7.8) | 29.9 (8.4) | 40.1 (7.1) | 14.6 (5.7)

2. Secondary Outcome: MATRICS
Description: MATRICS Consensus Cognitive Battery Performance: This is a standardized neurocognitive battery that assesses performance in 7 domains of neurocognition. Primary data are recorded based on normalized T-scores; a separate score is provided for each domain, and a Comprehensive score (Primary measure here) is also calculated across domains. Possible T-score range is 0 - 100; higher score reflects better performance.
Time Frame: approx 1 hour
Measure: Mean (Standard Error); unit: standardized T-score
Arm/Group | Subjects With Schizophrenia: Placebo 1st, Then 10 mg Memantine | Healthy Subjects: Placebo 1st, Then 10 mg Memantine | Subjects With Schizophrenia: 10 mg Memantine 1st, Then Placebo | Healthy Subjects: 10 mg Memantine 1st, Then Placebo | Subjects With Schizophrenia: Placebo 1st, Then 20 mg Memantine | Healthy Subjects: Placebo 1st, Then 20 mg Memantine | Subjects With Schizophrenia: 20 mg Memantine 1st, Then Placebo | Healthy Subjects: 20 mg Memantine 1st, Then Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10
standardized T-score
  Placebo | 40.4 (3.8) | 53.4 (2.3) | 41.1 (3.8) | 56.3 (2.4) | 34.2 (4.4) | 48.6 (4.3) | 37.7 (4.6) | 66.6 (2.0)
  Memantine | 44.6 (4.5) | 60.2 (2.7) | 34.3 (3.3) | 56.6 (6.6) | 35.8 (4.8) | 53.7 (5.8) | 31.0 (4.5) | 57.6 (1.9)

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Memantine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/80 | 0/80
Serious Adverse Events (participants affected / at risk) | 0/80 | 0/80
Other Adverse Events (participants affected / at risk) | 0/80 | 0/80

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-08-17): https://cdn.clinicaltrials.gov/large-docs/97/NCT01555697/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-17): https://cdn.clinicaltrials.gov/large-docs/97/NCT01555697/SAP_001.pdf